CLINICAL TRIAL: NCT03404505
Title: Effects of a Short-term Parent Mediated Social Training on Developmental Trajectories in Infants
Acronym: IA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Rebecca Landa, Principal Investigator, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00065698; R21DC015846 (NIH)
Record Dates: First submitted 2017-10-19; First posted 2018-01-19 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Younger Sibling of Child With Autism Spectrum Disorder; Signs of Developmental Delay; Signs of Communication Delay; Signs of Social Delay
Keywords: infant; play; parents

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infant Achievements (Experimental): Families randomized to the IA condition will receive 17 in-home sessions. These include a one-time start up session followed by twice-weekly visits in which they will be coached on how to implement the IA strategies. Families will receive a set of developmentally appropriate toys.
  Interventions: Behavioral: Infant Achievements
- Caregiver Education (Experimental): In this condition, parents will receive 17 sessions with a trained study team member focused on promoting child development and well-being. Sessions include a one-time start-up visit followed by one in-home visit and one phone contact per week. Families will receive a set of developmentally appropriate toys.
  Interventions: Behavioral: Caregiver Education (CE)

INTERVENTIONS:
Behavioral: Infant Achievements — Play-based intervention for caregivers and infants. The efficacy of the Infant Achievements intervention for improving communication and social behavior in infants who are at risk for communication, social, or developmental delay.
  Arms: Infant Achievements
Behavioral: Caregiver Education (CE) — Parents in the CE group will be taught about child development and well-being in their home, weekly, with a weekly follow-up phone call by trained research staff.
  Arms: Caregiver Education

SUMMARY:
This study is being done to examine the feasibility and impact of the Infant Achievements caregiver coaching treatment on caregiver child-engagement strategies used during play with their infant. The investigators will examine effects on infants' social and communication behavior. This randomized controlled trial will compare caregivers and infants in the Infant Achievements (IA) coaching group to caregivers and infants in the Caregiver Education (CE) no-coaching group. A total of 64 eligible participants (16 children plus their caregiver per group) will participate in the study.

DETAILED DESCRIPTION:
This study is being done to examine the feasibility and impact of the Infant Achievements caregiver coaching treatment on caregiver child-engagement strategies used during play with their infant. The investigators will examine effects on infants' social and communication behavior. This randomized controlled trial will compare caregivers and infants in the Infant Achievements (IA) coaching group to caregivers and infants in the Caregiver Education (CE) no-coaching group. A total of 64 eligible participants (16 children plus their caregiver per group) will participate in the study. Parents in the IA group will be coached, at home twice a week, to implement the intervention by trained research staff. Parents in the CE group will be taught about child development and well-being in their home, weekly, with a weekly follow-up phone call by trained research staff. In both groups: Videotaped caregiver-child interaction data will be gathered in the home. Baseline, post-treatment and follow-up measures will also be collected at the investigators' child development research center.

Families with children between the ages of 8 and 12 months with developmental concerns may be eligible to participate. Developmental concerns are defined as infrequent production of specific communication or social behaviors, or in immature or qualitatively atypical forms. These concerns will be documented via the Autism Observation Scale for Infants, Communication and Symbolic Behavior Scale (CSBS) Infant-Toddler Checklist, and/or Mullen Scales of Early Learning. Recruitment will occur from the Kennedy Krieger Institute (KKI), community agencies, and community events. Recruitment flyers will be distributed within those programs. In addition, a social media blurb will be placed on the KKI and other relevant groups' Facebook pages, KKI Center for Autism and Related Disorders newsletter, KKI websites, and may be sent to relevant local newsletters/magazines for families of young children.

ELIGIBILITY:
Inclusion Criteria:

* Child participants must be between the ages of 8 months and 12 months at the beginning of the study.
* Family must speak English at least 75% in the home.
* Children must receive an AOSI concern score ≥7 OR
* a T-score of ≤39 on either the Mullen Receptive Language or Expressive Language subscale. OR
* Score in the Concern range on either the Composite or Total Score of the parent-completed Communication and Symbolic Behavior Scales Developmental Profile (CSBS DP) Infant-Toddler Checklist.

Exclusion Criteria:

* History of head injury, seizure disorder, severe aggression or self-injurious behavior, prenatal illicit drug or excessive alcohol exposure.
* Any hearing or visual impairment
* Any severe birth trauma
* Any birth defects or genetic disorders
* Gestational age < 35 weeks and/or Birth weight less than 1,500g
* Cannot be living in foster care.
* Location of in-home visits >35 miles of the Center for Autism and Related Disorders

Ages: 8 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Change in parent behavior during the Parent-Child Play Sample | Change from behavior at Baseline to behavior at 8 weeks post-baseline, and from Baseline to 8 weeks post-intervention
  This measure is a natural observation of parent and child unstructured playing, and will be used to assess change in caregiver's use of child-responsive engagement strategies
Change in child communication and social engagement sample during the Parent-Child Play Sample | Change from behavior at Baseline to behavior at 8 weeks post-baseline, and from Baseline to 8 weeks post-intervention
  This outcome will be coded from the Parent-Child Play Sample

SECONDARY OUTCOMES:
Change in scores on the Mullen Scales of Early Learning Receptive and Expressive Language Raw Scores | Change from Baseline to 8 weeks post-baseline and from Baseline to 8 weeks post-intervention
  Receptive Language score (score range 0-48); Expressive Language Score (score range 0-50); higher scores indicate better outcome for both scales
Change in scores on the MacArthur-Bates Communication Development Inventory | Change from Baseline to 8 weeks post-baseline and from Baseline to 8 weeks post-intervention
  Number of words understood (range 0-396); Number of words produced (0-396); Total actions & gestures (0-63); higher scores indicate better outcomes for all scales
Change in scores on the CSBS Behavior Sample | Change from Baseline to 8 weeks post-baseline and from Baseline to 8 weeks post-intervention
  Frequency of initiation of joint attention; frequency of communicative consonants (range 0-6), gestures (range 0-6) and words (range (0-6); higher scores indicate greater outcome on all scales

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Landa, PhD, CCC-SLP, Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landa RJ, Reetzke R, Hess CR. Infant Achievements Intervention Improves Caregiver Implementation Fidelity and Infant Social Communication Outcomes: A Preliminary Randomized Clinical Trial. Autism Res. 2025 May;18(5):1104-1116. doi: 10.1002/aur.70051. Epub 2025 May 2. PMID 40318004